CLINICAL TRIAL: NCT03816579
Title: A Meal-based Comparison of Protein Quality, Complementary Proteins and Muscle Anabolism
Acronym: MAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 18-0147
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2020-12

CONDITIONS: Protein; Diet; Skeletal Muscle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PRO-A (Experimental): Beef protein
  Interventions: Other: PRO-A
- PRO-B (Experimental): Complementary proteins at each meal
  Interventions: Other: PRO-B
- PRO-C (Experimental): Complementary proteins over 24 hours
  Interventions: Other: PRO-C
- CON (No Intervention): Low protein (<5 g) meal

INTERVENTIONS:
Other: PRO-A — 30 g of beef protein will be consumed at each meal
  Arms: PRO-A
Other: PRO-B — 30 g of complementary proteins will be consumed at each meal
  Arms: PRO-B
Other: PRO-C — 30 g of complementary proteins will be consumed over 24 hours
  Arms: PRO-C

SUMMARY:
To highlight the importance of protein quality rather than the total protein content of a meal, the investigators will demonstrate that unlike high quality proteins, a single meal containing 30 g of an incomplete protein source does not stimulate skeletal muscle protein synthesis. Secondly, the investigators will directly challenge a prevalent, but untested, assertion that has the potential to negatively impact health. The goal is to demonstrate that complementary plant-proteins (i.e., two or more incomplete protein sources) must be consumed at the same meal to stimulate protein synthesis.

DETAILED DESCRIPTION:
The investigators will test the following hypotheses in middle-aged men and women (45-60) years old using a randomized, cross over design. All study objectives will be met concurrently:

1. Meals containing 30 g of high quality, predominantly beef-protein (PRO-A) will stimulate acute (i.e., single meal response) and 24 h skeletal muscle protein synthesis [confirmatory hypothesis]
2. Meals containing 30 g of complementary plant-based proteins (PRO-B: complete essential amino acid profile at each meal) will stimulate acute and 24 h skeletal muscle protein synthesis, but to a lesser extent than beef-protein.
3. A single meal containing 30 g of an incomplete plant-based protein source (PRO-C: lacking one essential amino acid) will fail to acutely stimulate skeletal muscle protein synthesis
4. Meals containing 30 g of plant-based protein that are incomplete at each separate meal, but complementary over a 24 h period, will fail to stimulate 24 h skeletal muscle protein synthesis.
5. Beef-and plant-based meals will have a similar effect on satiety and 24 h blood glucose [descriptive]

If these hypotheses are correct, the investigators will demonstrate that meals containing a moderate amount of high quality protein, such as beef, are an efficient and effective way to augment a largely plant based diet and stimulate skeletal muscle protein synthesis - a prerequisite for outcomes related to physical function, performance, successful aging and metabolic health.

ELIGIBILITY:
Inclusion Criteria:

1. All races and ethnic backgrounds
2. Men and women, age 45-60 years
3. Generally healthy (see exclusion criteria)
4. Able and willing to provide informed consent
5. Ability to speak and read English (* the study procedures, e.g., muscle biopsy, duration of each acute study, e.g. overnight stay; and multiple dietary questionnaires require sound written and spoken English)

Exclusion Criteria:

1. Sarcopenia (defined by: European Working Group on Sarcopenia in Older People, EWGSOP (44))
2. Clinically significant heart disease (e.g. New York Heart Classification greater than grade II; ischemia)
3. Peripheral vascular disease
4. Pulmonary disease
5. History of systemic or pulmonary embolus
6. Uncontrolled blood pressure (systolic BP>170, diastolic BP>95 mmHg)
7. Impaired renal function (creatinine >1.5 mg/dl)
8. Anemia (hematocrit <33)
9. Untreated thyroid disease (abnormal TSH)
10. A recent history (<12 months) of GI bleed
11. Diabetes mellitus or other untreated endocrine or metabolic disease
12. Electrolyte abnormalities
13. Any history of stroke, hypo- or hyper-coagulation disorders
14. Recent (3 years) treated cancer other than basal cell carcinoma
15. Systemic steroids, anabolic steroids, growth hormone or immunosuppressant use within 12 months
16. Recent (6 months) adherence to a weight-loss or weight-gain diet
17. Weight change of 5% or more in previous 6 months
18. Body mass index >30 or excess body fat that compromises muscle biopsy collection
19. Body mass index <20 or recent history (<12 month) of disordered eating
20. Dietary preferences or practices that preclude the consumption of the study meals
21. Acute infectious disease or chronic infection
22. Alcohol or drug abuse
23. Any other condition or event considered exclusionary by study physician
24. Pregnancy

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Acute muscle protein synthesis: PRO-A | 3 hours after consuming meal
  Muscle protein synthesis response to PRO-A breakfast meal (%/h)
Acute muscle protein synthesis: PRO-B | 3 hours after consuming meal
  Muscle protein synthesis response to PRO-B breakfast meal (%/h)
Acute muscle protein synthesis: PRO-C | 3 hours after consuming meal
  Muscle protein synthesis response to PRO-C breakfast meal (%/h)
Acute muscle protein synthesis: CON | 3 hours after consuming meal
  Muscle protein synthesis response to CON breakfast meal (%/hour)
24-hour muscle protein synthesis: PRO-A | Approximately 24 hours
  Muscle protein synthesis response to PRO-A diet over 24 hours (%/hour)
24-hour muscle protein synthesis: PRO-B | Approximately 24 hours
  Muscle protein synthesis response to PRO-B diet over 24 hours (%/hour)
24-hour muscle protein synthesis: PRO-C | Approximately 24 hours
  Muscle protein synthesis response to PRO-C diet over 24 hours (%/hour)
Blood amino acid response to diet: PRO-A | Approximately 5 hours
  Blood samples will be drawn to measure amino acid concentrations response to PRO-A breakfast (µmol/L)
Blood amino acid response to diet: PRO-B | Approximately 5 hours
  Blood samples will be drawn to measure amino acid concentrations response to PRO-B breakfast (µmol/L)
Blood amino acid response to diet: PRO-C | Approximately 5 hours
  Blood samples will be drawn to measure amino acid concentrations response to PRO-B C breakfast (µmol/L)
Blood amino acid response to diet: CON | Approximately 5 hours
  Blood samples will be drawn to measure amino acid concentrations response to CON breakfast (µmol/L)

SECONDARY OUTCOMES:
Blood glucose response to diet: PRO-A | Approximately 24 hours
  Blood samples will be drawn to measure blood glucose response to PRO-A diet (mg/dl)
Blood glucose response to diet: PRO-B | Approximately 24 hours
  Blood samples will be drawn to measure blood glucose response to PRO-B diet (mg/dl)
Blood glucose response to diet: PRO-C | Approximately 24 hours
  Blood samples will be drawn to measure blood glucose response to PRO-C diet (mg/dl)
Blood glucose response to diet: CON | Approximately 5 hours
  Blood samples will be drawn to measure blood glucose response to CON breakfast meal (mg/dl)
Appetite and Hedonic Questionnaire: PRO-A | Approximately 8 hours
  Questionnaires will be given to assess hunger, fullness, desire to eat, thirst, desire to eat something sweet, desire to eat something salty, desire to eat something savory, sleepiness, physical energy, mental energy, and nausea in response to PRO-A diet. All outcomes are scored individually on a 10 pt visual analog scale using "not at all" being 0 and "extremely" being a 10.
Appetite and Hedonic Questionnaire: PRO-B | Approximately 8 hours
  Questionnaires will be given to assess hunger, fullness, desire to eat, thirst, desire to eat something sweet, desire to eat something salty, desire to eat something savory, sleepiness, physical energy, mental energy, and nausea in response to PRO-B diet. All outcomes are scored individually on a 10 pt visual analog scale using "not at all" being 0 and "extremely" being a 10.
Appetite and Hedonic Questionnaire: PRO-C | Approximately 8 hours
  Questionnaires will be given to assess hunger, fullness, desire to eat, thirst, desire to eat something sweet, desire to eat something salty, desire to eat something savory, sleepiness, physical energy, mental energy, and nausea in response to PRO-C diet. All outcomes are scored individually on a 10 pt visual analog scale using "not at all" being 0 and "extremely" being a 10.
Appetite and Hedonic Questionnaire: CON | Approximately 5 hours
  Questionnaires will be given to assess hunger, fullness, desire to eat, thirst, desire to eat something sweet, desire to eat something salty, desire to eat something savory, sleepiness, physical energy, mental energy, and nausea in response to CON diet. All outcomes are scored individually on a 10 pt visual analog scale using "not at all" being 0 and "extremely" being a 10.
3 day dietary record: PRO-A | Approximately 36 hours
  Diet records will be collected and analyzed with ASA24 to assess habitual energy intake the week prior to PRO-A study visit
3 day dietary record: PRO-B | Approximately 36 hours
  Diet records will be collected and analyzed with ASA24 to assess habitual energy intake the week prior to PRO-B study visit
3 day dietary record: PRO-C | Approximately 36 hours
  Diet records will be collected and analyzed with ASA24 to assess habitual energy intake the week prior to PRO-C study visit
3 day dietary record: CON | Approximately 36 hours
  Diet records will be collected and analyzed with ASA24 to assess habitual energy intake the week prior to CON study visit
Palatability Questionnaire:PRO-A | Approximately 8 hours
  Questionnaires will be given to assess palatability of the PRO-A diet. Outcomes include the participants ranking of the food appearance, aroma intensity, aroma, flavor intensity, flavor, texture and overall appeal of the food. A 10 pt visual analog scale will be used to assess the subject's response with 0 being "extremely dislike", 5 being "neither like nor dislike" and 10 being "extremely like".
Palatability Questionnaire:PRO-B | Approximately 8 hours
  Questionnaires will be given to assess palatability of the PRO-B diet. Outcomes include the participants ranking of the food appearance, aroma intensity, aroma, flavor intensity, flavor, texture and overall appeal of the food. A 10 pt visual analog scale will be used to assess the subject's response with 0 being "extremely dislike", 5 being "neither like nor dislike" and 10 being "extremely like".
Palatability Questionnaire:PRO-C | Approximately 8 hours
  Questionnaires will be given to assess palatability of the PRO-C diet. Outcomes include the participants ranking of the food appearance, aroma intensity, aroma, flavor intensity, flavor, texture and overall appeal of the food. A 10 pt visual analog scale will be used to assess the subject's response with 0 being "extremely dislike", 5 being "neither like nor dislike" and 10 being "extremely like".
Palatability Questionnaire:CON | Approximately 5 hours
  Questionnaires will be given to assess palatability of the CON diet. Outcomes include the participants ranking of the food appearance, aroma intensity, aroma, flavor intensity, flavor, texture and overall appeal of the food. A 10 pt visual analog scale will be used to assess the subject's response with 0 being "extremely dislike", 5 being "neither like nor dislike" and 10 being "extremely like".

CONTACTS AND LOCATIONS:
Overall Officials: Doug Paddon-Jones, PhD, Principal Investigator — University of Texas
Locations (1):
- Unversity of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arentson-Lantz EJ, Von Ruff Z, Connolly G, Albano F, Kilroe SP, Wacher A, Campbell WW, Paddon-Jones D. Meals Containing Equivalent Total Protein from Foods Providing Complete, Complementary, or Incomplete Essential Amino Acid Profiles do not Differentially Affect 24-h Skeletal Muscle Protein Synthesis in Healthy, Middle-Aged Women. J Nutr. 2024 Dec;154(12):3626-3638. doi: 10.1016/j.tjnut.2024.10.010. Epub 2024 Oct 11. PMID 39396760